CLINICAL TRIAL: NCT00710593
Title: Immunogenicity, Safety, Tolerability, and Behavioral Consequences of an HPV-6, -11, -16, -18 Vaccine in HIV-Infected Young Women
Brief Title: Impact of a Human Papilloma Virus (HPV) Vaccine in HIV-Infected Young Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATN 064
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-04

CONDITIONS: HIV Infection
Keywords: Highly-active antiretroviral therapy; Human papillomavirus; HPV vaccine
MeSH Terms: conditions — HIV Infections | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: HAART naive or no HAART in past 6 months (Active Comparator): Participants who are ART naïve or, if ART-exposed, have not received highly active antiretroviral therapy (HAART) for at least the six months prior to study entry. All subjects will receive three doses of the HPV-6, -11, -16, -18 vaccine at the recommended dose and schedule (Day 0, Week 8, and Week 24).
  Interventions: Biological: HPV vaccine for strains -6, -11, -16, and -18
- B: HAART atleast 6 months/ 2 viral loads <400 in last 6 months (Active Comparator): Participants who have been receiving highly active antiretroviral therapy (HAART) for at least six months at the time of study entry, with two HIV-1 RNA plasma viral loads < 400 copies/ml on two previous clinical visits within the 6 months prior to study entry. All subjects will receive three doses of the HPV-6, -11, -16, -18 vaccine at the recommended dose and schedule (Day 0, Week 8, and Week 24).
  Interventions: Biological: HPV vaccine for strains -6, -11, -16, and -18

INTERVENTIONS:
Biological: HPV vaccine for strains -6, -11, -16, and -18 — All subjects will receive three doses of the HPV-6, -11, -16, -18 vaccine at the recommended dose and schedule (Day 0, Week 8, and Week 24).

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, safety, tolerability, and behavioral impact of an HPV-6, -11, -16, -18 vaccine in HIV-infected young women.

ELIGIBILITY:
Inclusion Criteria:

* Young women age 16 years and 0 days to 23 years and 364 days
* HIV-infection after the age of 9 years as documented by a positive result on any of the following licensed tests: any antibody test confirmed by Western blot, HIV-1 culture, HIV-1 DNA polymerase chain reaction (PCR), or plasma HIV-1 RNA > 1,000 copies/ml
* HIV treatment history that falls in one of the following categories:

Group A: ART naïve or if ART-exposed, has not received HAART for at least the six months prior to study entry Group B: Has been receiving HAART for at least six months at the time of study entry, with two HIV-1 RNA plasma viral loads < 400 copies/ml on two previous clinical visits within the 6 months prior to study entry

* Willingness to avoid pregnancy from study entry through the Week 28 visit for subjects of child-bearing potential, i.e., use of at least one barrier or hormonal method; e.g., condoms, Depo-Provera, oral contraceptive pills, etc. Subjects on antiretroviral (ARV) medications must use a barrier contraceptive method because ARV medications can make hormonal birth control less effective.
* Anticipated ability and willingness to complete all study vaccines and evaluations
* Ability and willingness to participate in the study by providing written informed consent

Exclusion Criteria:

* History of any prior vaccination with an HPV vaccine
* Active anogenital warts within three months prior to study entry) or history of cervical intraepithelial neoplasia (CIN) 2/3 (ever, must be documented by colposcopy)
* Previous allergic reaction to any constituents of the HPV vaccine
* Pregnancy
* Active substance use or dependence that, in the opinion of the site personnel, would interfere with adherence to the study
* Active opportunistic infection or current treatment for known or suspected active serious bacterial infection at the time of study entry
* Presence of any known > Grade 3 clinical or laboratory toxicity at the time of study entry (per the Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) Toxicity Tables, see ATN MOGO) with the exception of isolated Grade 3 serum total hyperbilirubinemia that is considered due to atazanavir (see Section 9.6 for definition of isolated total hyperbilirubinemia).
* Receipt of any routine vaccine within four weeks prior to study entry
* Receipt of any immune globulin or plasma product within six months prior study entry
* Receipt of any blood product or transfusion, other than immune globulin or plasma as noted above, within four weeks prior to study entry
* Receipt of any restricted medication listed in Section 5.3.2 within the four weeks preceding study entry
* Receipt of any other disallowed medication listed in Section 5.3.3 within the three months preceding study entry
* Thrombocytopenia or coagulation disorder that would contraindicate intramuscular injection
* Anticipation of long-term systemic corticosteroid therapy (more than 10 mg/day of prednisone or equivalent for > 2 consecutive weeks)
* Receipt of corticosteroid therapy at the above dose and duration within 3 months preceding study entry. Use of non-steroidal anti-inflammatory agents and inhaled or topical corticosteroids are not exclusion criteria
* Known or suspected disease of the immune system (other than HIV), i.e., malignancy, current or prior treatment for malignancy
* If other serious, acute or chronic medical or surgical conditions or contraindications are present during screening, the Protocol Team must be consulted to determine whether enrollment may interfere with the evaluation of the protocol objectives and for permission to proceed with the enrollment

Ages: 16 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A. Kahn, M.D., M.P.H., Study Chair — Adolescent Trials Network; Kathleen Squires, M.D., Study Chair — Adolescent Trials Network
Locations (14):
- United States (13):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Childrens Diagnostic & Treatment Center, Fort Lauderdale, Florida
  - University of Miami School of Medicine, Miami, Florida
  - USF College of Medicine, Tampa, Florida
  - Ruth M Rothstein CORE Center/ John H Stroger Jr Hospital, Chicago, Illinois
  - Childrens Memorial Hospital, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St Jude Childrens Research Hospital, Memphis, Tennessee
- University of Puerto Rico, Medical Sciences Campus, San Juan, Puerto Rico

REFERENCES:
- [Result] Kahn JA, Xu J, Zimet GD, Liu N, Gonin R, Dillard ME, Squires K; Adolescent Trials Network for HIV/AIDS Interventions. Risk perceptions after human papillomavirus vaccination in HIV-infected adolescents and young adult women. J Adolesc Health. 2012 May;50(5):464-70. doi: 10.1016/j.jadohealth.2011.09.005. Epub 2011 Nov 4. PMID 22525109
- [Result] Kahn JA, Burk RD, Squires KE, Kapogiannis BG, Rudy B, Xu J, Gonin R, Liu N, Worrell C, Wilson CM. Prevalence and risk factors for HPV in HIV-positive young women receiving their first HPV vaccination. J Acquir Immune Defic Syndr. 2012 Nov 1;61(3):390-9. doi: 10.1097/QAI.0b013e3182676fe3. PMID 22820809
- [Result] Kahn JA, Xu J, Kapogiannis BG, Rudy B, Gonin R, Liu N, Wilson CM, Worrell C, Squires KE. Immunogenicity and safety of the human papillomavirus 6, 11, 16, 18 vaccine in HIV-infected young women. Clin Infect Dis. 2013 Sep;57(5):735-44. doi: 10.1093/cid/cit319. Epub 2013 May 10. PMID 23667266
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — https://www.atnonline.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between 2008 and 2011 at Adolescent Trials Network for HIV/AIDS Interventions (ATN) clinical sites.
Groups:
- ART/HAART NAIVE: Participants who are antiretroviral (ART) naïve or, if ART-exposed, have not received highly active antiretroviral therapy (HAART) for at least the six months prior to study entry.
- HAART: Participants who have been receiving highly active antiretroviral therapy (HAART) for at least six months at the time of study entry, with two HIV-1 RNA plasma viral loads < 400 copies/ml on two previous clinical visits within the 6 months prior to study entry.
Period: Overall Study
Arm/Group | ART/HAART NAIVE | HAART
Started | 69 | 30
Completed | 54 (54 completed study and vaccine. 6 did not receive all vaccine, but completed all study visits.) | 25 (25 completed study and vaccine. 2 did not receive all vaccine, but completed all study visits.)
Not Completed | 15 | 5
Not completed — Incarceration | 1 | 0
Not completed — Unable to complete Wk 48 within window | 2 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Moved out of area | 1 | 0
Not completed — Failure to adhere or complete study eval | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Prem disc vaccine, completed all visits | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group A: Participants who are antiretroviral (ART) naïve or, if ART-exposed, have not received highly active antiretroviral therapy(HAART) for at least the six months prior to study entry.
- Group B: Participants who have been receiving highly active retroviral therapy (HAART) for at least six months at the time of study entry, with two HIV-1 RNA plasma viral loads < 400 copies/ml on two previous clinical visits within the 6 months prior to study entry.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 69 | 30 | 99
Age, Customized [Number; unit: Participants]
  < 20 years | 16 | 6 | 22
  > = 20 years | 53 | 24 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 30 | 99
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 63 | 29 | 92
  Puerto Rico | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: HPV-6 Antibody Level (Geometric Mean Titer of HPV-6)
Description: The outcome measure for the primary objective is immunogenicity as measured by the GMT of HPV-6, -11, -16, -18 vaccine four weeks after the administration of vaccine dose #3, measured as a continuous variable. Vaccine dose # 3 was administered at Week 24.
Time Frame: Week 28
Population: Subjects received the 3rd dose of vaccine and were both Human Papilloma Virus (HPV) Deoxyribonucleic Acid (DNA) negative and HPV-6 sero-negative at baseline (BL).
Measure: Geometric Mean (Standard Deviation); unit: Milli-Merck units/milliliter (mMU/mL)
Groups:
- All Study Participants Compared w/ Historical Comparison Group: This is a one sample test. This one-arm comparison compared the mean geometric mean titers (GMTs) to HPV-6 four weeks post vaccine dose #3 in study subjects with cluster of differentiation 4 (CD4+) T-cell counts > 350 mm3 with a null value: the mean GMT of HIV-negative and HPV vaccinated subjects in industry-sponsored trials.
  Comparing data collected from this study to results from a historical comparison group is part of the protocol design.
Arm/Group | All Study Participants Compared w/ Historical Comparison Group
Number analyzed (Participants) | 40
Milli-Merck units/milliliter (mMU/mL) | 738.9 (908.7)

2. Secondary Outcome: Immunogenicity of the HPV-6, -11, -16, -18 Vaccine Four Weeks After Vaccine Dose #3 as Measured as a Binary Variable (Responder vs. Non-responder) for HPV-6
Description: Subjects who had a greater than or equal to (>=) 20 Milli-Merck units (mMU)/milliliter (mL) response were classified as responders; subjects who had a less than (<) 20 mMU/mL response were classified as non-responders.
Time Frame: Week 28
Population: Subjects had received third dose of vaccination who were both Human Papilloma Virus (HPV) Deoxyribonucleic Acid (DNA) negative and HPV Sero-Negative at baseline.
Measure: Number; unit: participants
Groups:
- All Study Participants Compared w/ Historical Comparison Group: The results are reported for all participants in both Group A and Group B.
Arm/Group | All Study Participants Compared w/ Historical Comparison Group
Number analyzed (Participants) | 40
participants
  Responder | 39
  Non-Responder | 1
Statistical Analysis 1: Comparison: All Study Participants Compared w/ Historical Comparison Group; Historical comparison group can be referenced in: Villa et al. Immunologic responses following administration of a vaccine targeting human papillomavirus Types 6, 11, 16, and 18; Vaccine 24 (2006):5571-5583. PMID 16753240; Test type: Superiority or Other; p = 0.1613, Fisher Exact; % of participants who were responders = 97.5, 95% CI 2-sided [86.8 to 99.9]

3. Secondary Outcome: Immunogenicity of the HPV-6, -11, -16, -18 Vaccine Four Weeks After Vaccine Dose #3 as Measured as a Binary Variable (Responder vs. Non-responder) for HPV-11
Description: Subjects who had a >= 16 mMU/mL were classified as responders; subjects who had a less than < 16 mMU/mL response were classified as non-responders.
Time Frame: Week 28
Population: Subjects had received third dose of vaccination who were both HPV DNA negative and HPV Sero-Negative at baseline.
Measure: Number; unit: participants
Arm/Group | All Study Participants Compared w/ Historical Comparison Group
Number analyzed (Participants) | 63
participants
  Responders | 61
  Non-Responders | 2
Statistical Analysis 1: Comparison: All Study Participants Compared w/ Historical Comparison Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0534, Fisher Exact; % of participants who were responders = 96.8, 95% CI 2-sided [89.0 to 99.9]

4. Secondary Outcome: Immunogenicity of the HPV-6, -11, -16, -18 Vaccine Four Weeks After Vaccine Dose #3 as Measured as a Binary Variable (Responder vs. Non-responder) for HPV-16
Description: Subjects who had a >= 20 mMU/mL were classified as responders; subjects who had a less than < 20 mMU/mL response were classified as non-responders.
Time Frame: Week 28
Population: Subjects had received third dose of vaccination who were both HPV DNA negative and HPV Sero-Negative at baseline.
Measure: Number; unit: participants
Arm/Group | All Study Participants Compared w/ Historical Comparison Group
Number analyzed (Participants) | 51
participants
  Responders | 49
  Non-Responders | 2
Statistical Analysis 1: Comparison: All Study Participants Compared w/ Historical Comparison Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0427, Fisher Exact; % of participants who were responders = 96.1, 95% CI 2-sided [86.5 to 99.5]

5. Secondary Outcome: Immunogenicity of the HPV-6, -11, -16, -18 Vaccine Four Weeks After Vaccine Dose #3 as Measured as a Binary Variable (Responder vs. Non-responder) for HPV-18
Description: Subjects who had a >= 24 mMU/mL were classified as responders; subjects who had a less than < 24 mMU/mL response were classified as non-responders.
Time Frame: Week 28
Population: Subjects had received third dose of vaccination who were both HPV DNA negative and HPV Sero-Negative at baseline.
Measure: Number; unit: participants
Arm/Group | All Study Participants Compared w/ Historical Comparison Group
Number analyzed (Participants) | 67
participants
  Responders | 62
  Non-Responders | 5
Statistical Analysis 1: Comparison: All Study Participants Compared w/ Historical Comparison Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0006, Fisher Exact; % of participants who were responders = 92.5, 95% CI 2-sided [83.4 to 97.5]

6. Secondary Outcome: Number of Participants With At Least One Adverse Event Possibly, Probably, or Definitely Related to Vaccine
Description: When a subject had at least one adverse event or sign/symptom during the study after doses 1, 2 or 3, and the event was possibly, probably, or definitely related to vaccine, this subject was considered to have had a vaccine-associated adverse event, sign and/or symptom.
Time Frame: Entry, Week 8, and Week 24
Population: Subjects who had at least one event that was possibly, probably, or definitely related to vaccine.
Measure: Number; unit: participants
Groups:
- All Study Participants: All study participants who were administered vaccine doses #1, 2, and/or 3.
Arm/Group | All Study Participants
Number analyzed (Participants) | 99
participants
  Group A: number analyzed (Participants) | 69
  Group A | 34
  Group B: number analyzed (Participants) | 30
  Group B | 14
Statistical Analysis 1: Comparison: All Study Participants; Test type: Superiority or Other; p = 0.8305, Chi-squared, Corrected — The p-value is to test the proportions of subjects with at least one event among Group A during the study at Entry, Week 8 and Week 24 after vaccine was administered; % of participants with at least 1 event = 49.3
Statistical Analysis 2: Comparison: All Study Participants; Test type: Superiority or Other; p = 0.8305, Chi-squared, Corrected — The p-value is to test the proportions of subjects with at least one event among Group B during the study at Entry, Week 8 and Week 24 after vaccine was administered; % of participants with at least 1 event = 46.7

7. Secondary Outcome: Persistence of Immunogenicity of the HPV-6, -11, -16, and -18 Vaccine 24 Weeks Post Vaccine Dose #3 as Measured by the Geometric Mean Titers (GMT) of HPV-6.
Description: Persistence of immunogenicity as measured by geometric mean titers (GMT) to HPV-6, -11, -16, -18 vaccine 24 weeks after the administration of vaccine dose #3, measured as a continuous variable. Vaccine dose #3 was administered at Week 24.
Time Frame: Week 48
Population: Subjects had received third dose of vaccination who were both HPV DNA negative and HPV sero-negative at baseline.
Measure: Geometric Mean (Standard Deviation); unit: Milli-Merck units/milliliter (mMU/mL)
Groups:
- All Study Participants: The results are reported for all study participants in both Group A and Group B.
Arm/Group | All Study Participants
Number analyzed (Participants) | 36
Milli-Merck units/milliliter (mMU/mL) | 311.9 (346.2)

8. Secondary Outcome: Persistence of Immunogenicity of the HPV-6, -11, -16, and -18 Vaccine 24 Weeks Post Vaccine Dose #3 as Measured by the Geometric Mean Titers (GMT) of HPV-11.
Description: Persistence of immunogenicity as measured by geometric mean titers (GMT) to HPV-6, -11, -16, -18 vaccine 24 weeks after the administration of vaccine dose #3, measured as a continuous variable. Vaccine dose # 3 was administered at Week 24
Time Frame: Week 48
Population: Subjects had received a third dose of vaccination who were both HPV DNA negative and HPV sero-negative at baseline.
Measure: Geometric Mean (Standard Deviation); unit: Milli-Merck units/milliliter (mMU/mL)
Groups:
- All Study Participants: The results are reported for participants in both Group A and Group B.
Arm/Group | All Study Participants
Number analyzed (Participants) | 56
Milli-Merck units/milliliter (mMU/mL) | 311.8 (448.7)

9. Secondary Outcome: Persistence of Immunogenicity of the HPV-6, -11, -16, and -18 Vaccine 24 Weeks Post Vaccine Dose #3 as Measured by the Geometric Mean Titers (GMT) of HPV-16.
Description: as for outcome 8
Time Frame: Week 48
Population: Subjects had received a third dose of vaccination who were both HPV DNA negative and HPV sero-negative at baseline.
Measure: Geometric Mean (Standard Deviation); unit: mMU/mL
Arm/Group | All Study Participants
Number analyzed (Participants) | 48
mMU/mL | 992.5 (1471.0)

10. Secondary Outcome: Persistence of Immunogenicity of the HPV-6, -11, -16, and -18 Vaccine 24 Weeks Post Vaccine Dose #3 as Measured by the Geometric Mean Titers (GMT) of HPV-18.
Description: as for outcome 8
Time Frame: Week 48
Population: Subjects had received a third dose of vaccination who were both HPV DNA negative and HPV sero-negative at baseline.
Measure: Geometric Mean (Standard Deviation); unit: mMU/mL
Arm/Group | All Study Participants
Number analyzed (Participants) | 62
mMU/mL | 175.3 (324.8)

11. Primary Outcome: HPV-11 Antibody Level (Geometric Mean Titer of HPV-11)
Description: The outcome measure for the primary objective is immunogenicity as measured by the GMTs of HPV-6, -11, -16, -18 vaccine four weeks after the administration of vaccine dose #3, measured as a continuous variable. Vaccine Dose #3 was administered at Week 24.
Time Frame: Week 28
Population: Subjects received the 3rd dose of vaccine and were both Human Papilloma Virus (HPV) Deoxyribonucleic Acid (DNA) negative and HPV-11 sero-negative at baseline (BL).
Measure: Geometric Mean (Standard Deviation); unit: mMU/mL
Groups:
- All Study Participants Compared w/ Historical Comparison Group: This is a one sample test. This one-arm comparison compared the mean geometric mean titers (GMTs) to HPV-11 four weeks post vaccine dose #3 in study subjects with cluster of differentiation 4 (CD4+) T-cell counts > 350 mm3 with a null value: the mean GMT of HIV-negative and HPV vaccinated subjects in industry-sponsored trials.
  Comparing data collected from this study to results from a historical comparison group is part of the protocol design.
Arm/Group | All Study Participants Compared w/ Historical Comparison Group
Number analyzed (Participants) | 63
mMU/mL | 896.0 (1132.1)

12. Primary Outcome: HPV-16 Antibody Level (Geometric Mean Titer of HPV-16)
Description: The outcome measure for the primary objective is immunogenicity as measured by the GMTs of HPV-6, -11, -16, -18 vaccine four weeks after the administration of vaccine dose #3, measured as a continuous variable. Vaccine dose # 3 was administered at Week 24.
Time Frame: Week 28
Population: Subjects received the 3rd dose of vaccine and were both Human Papilloma Virus (HPV) Deoxyribonucleic Acid (DNA) negative and HPV-16 sero-negative at baseline (BL).
Measure: Geometric Mean (Standard Deviation); unit: mMU/mL
Groups:
- All Study Participants Compared w/ Historical Comparison Group: This is a one sample test. This one-arm comparison compared the mean geometric mean titers (GMTs) to HPV-16 four weeks post vaccine dose #3 in study subjects with cluster of differentiation 4 (CD4+) T-cell counts > 350 mm3 with a null value: the mean GMT of HIV-negative and HPV vaccinated subjects in industry-sponsored trials.
  Comparing data collected from this study to results from a historical comparison group is part of the protocol design.
Arm/Group | All Study Participants Compared w/ Historical Comparison Group
Number analyzed (Participants) | 51
mMU/mL | 2961.1 (3376.8)

13. Primary Outcome: HPV-18 Antibody Level (Geometric Mean Titer of HPV-18)
Description: as for outcome 11
Time Frame: Week 28
Population: Subjects received the 3rd dose of vaccine and were both Human Papilloma Virus (HPV) Deoxyribonucleic Acid (DNA) negative and HPV-18 sero-negative at baseline (BL).
Measure: Geometric Mean (Standard Deviation); unit: mMU/mL
Groups:
- All Study Participants Compared w/ Historical Comparison Group: This is a one sample test. This one-arm comparison compared the mean geometric mean titers (GMTs) to HPV-18 four weeks post vaccine dose #3 in study subjects with cluster of differentiation 4 (CD4+) T-cell counts > 350 mm3 with a null value: the mean GMT of HIV-negative and HPV vaccinated subjects in industry-sponsored trials.
  Comparing data collected from this study to results from a historical comparison group is part of the protocol design.
Arm/Group | All Study Participants Compared w/ Historical Comparison Group
Number analyzed (Participants) | 67
mMU/mL | 576.5 (839.6)

14. Secondary Outcome: Acquisition of HPV-6 DNA by Study Group and Study Visit (Week 24).
Description: Type-specific HPV DNA among subjects who were both HPV DNA negative and HPV-6 sero-negative by study group and study visit at Week 24.
Time Frame: Week 24
Population: Subjects who were both Human Papilloma Virus (HPV) Deoxyribonucleic Acid (DNA) negative and HPV-6 sero-negative at Week 24. (The number of participants analyzed for this outcome differs from the number of participants in the Participant Flow Module.)
Measure: Number; unit: percentage of participants
Groups:
- Group A: Antiretroviral therapy (ART) naïve or if ART exposed, have not received highlight active antiretroviral (HAART) for at least the six months prior to study entry.
- Group B: Received highly active antiretroviral therapy (HAART) for at least six months at the time of study entry.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 26 | 12
percentage of participants
  Yes | 7.7 | 8.3
  No | 92.3 | 91.7
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority or Other; p = 1.000, Fisher Exact; P-value is from the Fisher's Exact test to compare the proportion of HPV positive between two study groups; Overall aquisition rate = 7.9

15. Secondary Outcome: Acquisition of HPV-11 DNA by Study Group and Study Visit (Week 24).
Description: Type-specific HPV DNA among subjects who were both HPV DNA negative and HPV-11 sero-negative by study group and study visit at Week 24.
Time Frame: Week 24
Population: Subjects who were both Human Papilloma Virus (HPV) Deoxyribonucleic Acid (DNA) negative and HPV-11 sero-negative at Week 24. (The number of participants analyzed for this outcome differs from the number of participants in the Participant Flow Module.)
Measure: Number; unit: percentage of participants
Groups:
- Group A: Participants who are ART naïve or, if ART-exposed, have not received highly active antiretroviral therapy (HAART) for at least the six months prior to study entry.
- Group B: Participants who have been receiving highly active antiretroviral therapy (HAART) for at least six months at the time of study entry, with two HIV-1 RNA plasma viral loads < 400 copies/ml on two previous clinical visits within the 6 months prior to study entry.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 43 | 19
percentage of participants
  Yes | 2.3 | 0.0
  No | 97.7 | 100.0
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value is from the Fisher's Exact test to compare the proportion of HPV positive between two study groups; Overall aquisition rate = 1.6

16. Secondary Outcome: Acquisition of HPV-16 DNA by Study Group and Study Visit (Week 24).
Description: Type-specific HPV DNA among subjects who were both HPV DNA negative and HPV-16 sero-negative by study group and study visit at Week 24.
Time Frame: Week 24
Population: Subjects who were both Human Papilloma Virus (HPV) Deoxyribonucleic Acid (DNA) negative and HPV-16 sero-negative for at Week 24. (The number of participants analyzed for this outcome differs from the number of participants in the Participant Flow Module.)
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 36 | 15
percentage of participants
  Yes | 2.8 | 0.0
  No | 97.2 | 100.0
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value is from the Fisher's Exact test to compare the proportion of HPV positive between two study groups; Overall aquisition rate = 2.0

17. Secondary Outcome: Acquisition of HPV-18 DNA by Study Group and Study Visit (Week 24).
Description: Type-specific HPV DNA among subjects who were both HPV DNA negative and HPV-18 sero-negative by study group and study visit at Week 24.
Time Frame: Week 24
Population: Subjects who were both Human Papilloma Virus (HPV) Deoxyribonucleic Acid (DNA) negative and HPV-18 sero-negative at Week 24. (The number of participants analyzed for this outcome differs from the number of participants in the Participant Flow Module.)
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 49 | 18
percentage of participants
  Yes | 4.1 | 5.6
  No | 95.9 | 94.4
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value is from the Fisher's Exact test to compare the proportion of HPV positive between two study groups; Overall aquisition rate = 4.5

18. Secondary Outcome: Acquisition of HPV-6 DNA by Study Group and Study Visit (Week 48).
Description: Type-specific HPV DNA among subjects who were both HPV DNA negative and HPV sero-negative by study group and study visit at Week 48.
Time Frame: Week 48
Measure: Number; unit: percentage of participants
Groups:
- Group A: Participants who are ART naïve or, if ART-exposed, have not received highly active antiretroviral therapy (HAART) for at least the six months prior to study entry. All subjects will receive three doses of the HPV-6, -11, -16, -18 vaccine at the recommended dose and schedule (Day 0, Week 8, and Week 24).
Arm/Group | Group A | Group B
Number analyzed (Participants) | 24 | 12
percentage of participants
  Yes | 8.3 | 8.3
  No | 91.7 | 91.7
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value is from the Fisher's Exact test to compare the proportion of HPV positive between two study groups; Overall aquisition rate = 8.3

19. Secondary Outcome: Acquisition of HPV-11 DNA by Study Group and Study Visit (Week 48).
Description: as for outcome 18
Time Frame: Week 48
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 39 | 17
percentage of participants
  Yes | 5.1 | 0.0
  No | 94.9 | 100.0
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value is from the Fisher's Exact test to compare the proportion of HPV positive between two study groups; Overall aquistion rate = 3.6

20. Secondary Outcome: Acquisition of HPV-16 DNA by Study Group and Study Visit (Week 48).
Description: as for outcome 18
Time Frame: Week 48
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 34 | 14
percentage of participants
  Yes | 5.9 | 7.1
  No | 94.1 | 92.9
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value is from the Fisher's Exact test to compare the proportion of HPV positive between two study groups; Overall aquisition rate = 6.3

21. Secondary Outcome: Acquisition of HPV-18 DNA by Study Group and Study Visit (Week 48).
Description: as for outcome 18
Time Frame: Week 48
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 46 | 16
percentage of participants
  Yes | 8.7 | 6.3
  No | 91.3 | 93.8
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value is from the Fisher's Exact test to compare the proportion of HPV positive between two study groups; Overall aquisition rate = 8.1

22. Secondary Outcome: Percentage of Participants Who Reported a Lower Need to Practice Safe Sex Following HPV Vaccination and the Percentage of Participants That Reported a Higher Need to Practice Safe Sex Following HPV Vaccination
Description: Participants' perceptions for the need to practice safe sex following HPV vaccination was measured using a safer sexual behaviors subscale, which was comprised of the following five questions:
  After getting vaccinated against HPV …
  1. You feel that condom use during sex is less necessary.
  2. You feel it is still just as important to have as few sexual partners as possible.
  3. You feel that it is less important to talk to your sex partners about safe sex.
  4. You think it is still just as important to use a condom every time you have sex.
  5. You will be less worried about having unprotected sex. Those who were categorized in the "lower need for safer sexual behaviors (NSSB)" group had a summary score that was less than the median and those in the "higher NSSB" group had a summary score that was equal to or higher than the median.
Time Frame: Week 48
Measure: Number; unit: percentage of participants
Groups:
- Lower NSSB: Lower NSSB is defined as participants who had a lower need for safer sexual behaviors (summary score is less than the median).
- Higher NSSB: Higher NSSB is defined as participants who had a higher need for safer sexual behaviors (summary score is equal to or greater than the median).
Arm/Group | Lower NSSB | Higher NSSB
Number analyzed (Participants) | 47 | 52
percentage of participants | 47.5 | 52.5
Statistical Analysis 1: Comparison: Lower NSSB vs Higher NSSB; Test type: Superiority or Other; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [1.02 to 1.1]

23. Secondary Outcome: Need for Safer Sexual Behaviors (NSSB) (Evaluated by Using the "12-item Knowledge About HPV and HPV Vaccine" Measure)
Description: To characterize young women's risk perceptions, sexual behaviors, and sexually transmitted infections (STI) diagnoses over the 48 weeks after initial vaccination, the relationship of baseline "12-item Knowledge About HPV and HPV Vaccine" measure was used to evaluate the need for safer sexual behaviors.
Time Frame: Week 48
Population: Total population analyzed was 99 participants. Percentage of participants reflects percentage of participants in both lower NSSB and higher NSSB.
Measure: Number; unit: percentage of participants
Arm/Group | Lower NSSB | Higher NSSB
Number analyzed (Participants) | 47 | 52
percentage of participants | 47.5 | 52.5
Statistical Analysis 1: Comparison: Lower NSSB vs Higher NSSB; Test type: Superiority or Other; p = 0.0012, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [1.0 to 1.1]

24. Secondary Outcome: Visit Compliance Via the Telephone Response System (TRS) Versus the Vaccine Report Card.
Description: Visit compliance is the total number of days participants actually called the TRS or completed the VRC divided by the total number of days expected to call the TRS or complete the VRC, multiplied by 100%.
Time Frame: Day 1 through Week 24
Measure: Mean (Standard Deviation); unit: percentage of days
Groups:
- Telephone Response System (TRS): Participants at sites randomized to the TRS called the TRS once a day to report any side effects they were experiencing.
- Vaccine Report Card (VRC): Participants at sites randomized to the VRC recorded any of their side effects. Participants were directed to call the clinical site staff or return to the clinic for evaluation if they were concerned about their signs or symptoms or if any symptoms appeared severe. Participants brought their VRC with them to all of their study visits. The completed cards were collected after all vaccine study visits were completed.
Arm/Group | Telephone Response System (TRS) | Vaccine Report Card (VRC)
Number analyzed (Participants) | 59 | 38
percentage of days | 51.3 (27.4) | 96.1 (14.0)
Statistical Analysis 1: Comparison: Telephone Response System (TRS) vs Vaccine Report Card (VRC); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

25. Secondary Outcome: Adverse Events (AE) Reported Among Participants Who Were Randomized to the Telephone Response System (TRS) or Vaccine Report Card (VRC).
Description: Rate of AEs is the total number of AEs divided by the total number of participants. The rate is not a percentage bur rather it could be above 1 or less than 1. This outcome measure looked at number of AEs reported, by grade; number of AEs > Grade 3 identified; and number of AEs > Grade 3 evaluated within 24 or 48 hours.
Time Frame: Day 1 through Week 24
Measure: Number; unit: AEs/Total Number of Participants
Groups:
- Vaccine Report Card (VRC): Participants at sites randomized to the VRC recorded any of their side effects.
Arm/Group | Telephone Response System (TRS) | Vaccine Report Card (VRC)
Number analyzed (Participants) | 59 | 38
AEs/Total Number of Participants
  Grade 1 | 0.93 | 1.37
  Grade 2 | 1.19 | 1.37
  Grade 3 | 0.07 | 0.08
  Grade 4 | 0.00 | 0.03
  Grade 3 or above identified after evaluation | 0.07 | 0.11
  Overall | 2.19 | 2.84

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: Participants were considered to have a vaccine-associated sign and/or symptom if they had at least one sign/symptom during the study after each vaccination, and the sign/symptom is possibly, probably, or definitely related to vaccine.
Groups:
- Group A: HAART naïve or, if HAART Exposed, Has Not Received HA: Participants who are ART naïve or, if ART-exposed, have not received HAART for at least the six months prior to study entry. All subjects will receive three doses of the HPV-6, -11, -16, -18 vaccine at the recommended dose and schedule (Day 0, Week 8, and Week 24).
- Group B: Has Been Receiving HAART for > 6 Months, With Two HIV: Participants who have been receiving HAART for at least six months at the time of study entry, with two HIV-1 RNA plasma viral loads < 400 copies/ml on two previous clinical visits within the 6 months prior to study entry. All subjects will receive three doses of the HPV-6, -11, -16, -18 vaccine at the recommended dose and schedule (Day 0, Week 8, and Week 24).
Arm/Group | Group A: HAART naïve or, if HAART Exposed, Has Not Received HA | Group B: Has Been Receiving HAART for > 6 Months, With Two HIV
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/30
Other Adverse Events (participants affected / at risk) | 34/69 | 14/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: HAART naïve or, if HAART Exposed, Has Not Received HA (N=69) | Group B: Has Been Receiving HAART for > 6 Months, With Two HIV (N=30)
Fever (General disorders) | 9 (18) | 3 (5)
Local reactions (General disorders) | 19 (25) | 7 (10) — Local reactions include pain and induration.
Systemic Reactions (General disorders) | 15 (35) | 9 (14) — Systemic reactions include: headache, fatigue, malaise, anorexia, arthralgia/myalgia and weakness.
Other Reactions (General disorders) | 5 (5) | 8 (9)

LIMITATIONS AND CAVEATS:
The small number of participants (99 started and 79 completed the study) limits generalizability of safety/tolerability data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Adolescent Medicine Trials Network (ATN) for HIV/AIDS Interventions Publication Policy outlines procedures for the development and review of abstracts, publications and presentations. The Adolescent Medicine Leadership Group (AMLG) retains custody of and primary rights to the data. Use of data must be approved by the protocol team and AMLG.